CLINICAL TRIAL: NCT02581384
Title: Stereotactic Body Radiotherapy (SBRT) for Pulmonary Metastases in Ewing Sarcoma, Rhabdomyosarcoma, and Wilms Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study closed primarily due to weak accrual, as well as study design limitations.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Karen J Marcus, MD FACR, Karen J Marcus, M.D., Boston Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-278
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Ewing Sarcoma; Rhabdomyosarcoma; Wilms Tumor; Osteosarcoma; Non-Rhabdomyosarcoma Soft Tissue Sarcoma, Nos; Renal Tumor; Rhabdoid Tumor; Clear Cell Renal Cell Carcinoma; Sarcoma; Sarcoma, Ewing; Soft Tissue Sarcoma
Keywords: Ewing Sarcoma; Rhabdomyosarcoma; Wilms Tumor; Rhabdomyosarcoma of Mediastinum; Ewing's Sarcoma Metastatic; Ewing Family of Tumors; Ewing's Tumor Metastatic; Osteosarcoma, Metastatic; Osteosarcoma in Children; Rhabdoid Tumor; Lung Metastasis; Radiation for Children; SBRT for children; Stereotactic Body Radiotherapy; Pulmonary Metastasis; Lung Metastasis in Children; Pulmonary Metastasis in Children; Comfort Care; Palliative Care
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Wilms Tumor; Osteosarcoma; Sarcoma; Carcinoma, Renal Cell; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive, Peripheral; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Cohort 1 Dose Level 1 [Phase I] (Experimental): Participants with Wilms tumors or other primary renal tumors. Stereotactic Body Radiotherapy (SBRT) Dose Levels for each target lesion are three 8 Gy fractions for 24 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 1 Dose Level 2 [Phase I] (Experimental): Participants with Wilms tumors or other primary renal tumors. SBRT Dose Levels for each target lesion are three 10 Gy fractions for 30 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 1 Dose Level 3 [Phase I] (Experimental): Participants with Wilms tumors or other primary renal tumors. SBRT Dose Levels for each target lesion are three 12 Gy fractions for 36 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 2 Dose Level 2 [Phase I] (Experimental): Participants with Ewing sarcoma or rhabdomyosarcoma. SBRT Dose Levels for each target lesion are three 10 Gy fractions for 30 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 2 Dose Level 3 [Phase I] (Experimental): Participants with Ewing sarcoma or rhabdomyosarcoma.SBRT Dose Levels for each target lesion are three 12 Gy fractions for 36 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)
- Cohort 2 Dose Level 2 [Phase II] (Experimental): Participants with Ewing sarcoma or rhabdomyosarcoma. SBRT Dose Levels for each target lesion are three 10 Gy fractions for 30 Gy total.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT)

SUMMARY:
This research study is studying stereotactic body radiotherapy (SBRT) as a possible treatment for lung relapse of Ewing sarcoma, rhabdomyosarcoma, osteosarcoma, non-rhabdomyosarcoma soft tissue sarcoma, Wilms tumor or other primary renal tumor (including clear cell and rhabdoid). SBRT is a form of targeted radiotherapy that can treat very small tumors using a few large doses.

DETAILED DESCRIPTION:
This research study is a Pilot Study, also known as a Phase I-II study, which means it is the first time investigators are examining this study intervention for patients with lung recurrence of Ewing sarcoma, rhabdomyosarcoma, osteosarcoma, nonrhabdomyosarcoma soft tissue sarcoma, Wilms tumor or other primary renal tumor (including clear cell and rhabdoid). This study tests the most appropriate dose, safety and efficacy of SBRT for the treatment of lung recurrence of these cancers in children. Standard radiotherapy is typically used to treat Ewing sarcoma and is used to treat lung recurrence. SBRT is being used to treat adults with small inoperable lung cancers; in such cases, SBRT has been shown to be effective and well-tolerated. SBRT is also used to treat bone metastases in adults and children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ewing sarcoma, rhabdomyosarcoma, osteosarcoma, non-rhabdomyosarcoma soft tissue sarcoma, Wilms tumor or other primary renal tumor (including clear cell and rhabdoid)
* Age ≤ 21 years;
* Must be capable of treatment without general anesthesia
* Lesion size 8 mm - 3 cm
* Subjects who have lesions within 2 cm of central structures, will be eligible on a case by-case basis
* Pulmonary metastases found at relapse (does not have to be first relapse); no more than 3 lesions per hemi-thorax will be treated but other lesions in the lung may be present
* Greater than 5 weeks from doxorubicin at the time of consent, with radiation to be initiated no less than 6 weeks from doxorubicin
* Informed consent/assent
* Life expectancy >3 months
* Pulmonary Function FEV1 ≥ 50% of predicted;
* Concurrent immunotherapy is allowed

Exclusion Criteria:

* Prior whole-lung or hemi-thorax irradiation of greater than 12 Gy received less than 6 months prior to consent (focal radiotherapy to the thorax is not an exclusion)
* Lesion larger than 3 cm in diameter
* Patients for whom surgery would be deemed appropriate rather than radiotherapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Marcus, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu KX, Chen YH, Kozono D, Mak RH, Boyle PJ, Janeway KA, Mullen EA, Marcus KJ. Phase I/II Study of Stereotactic Body Radiation Therapy for Pulmonary Metastases in Pediatric Patients. Adv Radiat Oncol. 2020 Sep 23;5(6):1267-1273. doi: 10.1016/j.adro.2020.09.004. eCollection 2020 Nov-Dec. PMID 33305087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2017 to December 2018. No participants were in enrolled in Cohort 1 Dose Level 1 [Phase I], Cohort 1 Dose Level 2 [Phase I], Cohort 1 Dose Level 3 [Phase I], and Cohort 2 Dose Level 3 [Phase I]
Groups:
- Cohort 2 Dose Level 2 [Phase I]; Cohort 2 Dose Level 2 [Phase II]: Participants with Ewing sarcoma or rhabdomyosarcoma. SBRT Dose Levels for each target lesion are three 10 Gy fractions for 30 Gy total.
  Stereotactic Body Radiotherapy (SBRT)
Period: Overall Study
Arm/Group | Cohort 2 Dose Level 2 [Phase I] | Cohort 2 Dose Level 2 [Phase II]
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2 Dose Level 2 [Phase I and II]: Participants with Ewing sarcoma or rhabdomyosarcoma. SBRT Dose Levels for each target lesion are three 10 Gy fractions for 30 Gy total.
  Stereotactic Body Radiotherapy (SBRT)
Arm/Group | Cohort 2 Dose Level 2 [Phase I and II]
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 12 [7 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
  Other | 1
  Unknown | 1
Primary Tumor Histologies [Count of Participants; unit: Participants]
  Ewing Sarcoma | 3
  Anaplastic Chordoma | 1
  Osteosarcoma | 1
Number of Lesions [Count of Participants; unit: Participants]
  Two Lesions | 3
  One Lesion | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity [Phase I]
Description: Dose Limiting Toxicities (DLT's) are toxicities experienced from start of therapy to 6 month. DLT's are assessed on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.
  DLTs are defined as follows:
  Grade 2 or higher toxicities:
  * Myelitis
  * Esophageal fistula, perforation, hemorrhage
  Grade 3 or higher toxicities considered to be a direct result of therapy:
  * Pneumonitis
  * Pericarditis, pericardial effusion
  * Esophageal necrosis, stenosis, ulcer
  * Dyspnea
  Grade 4 toxicities:
  * Esophagitis
  * Pericardial tamponade
  * Pulmonary toxicity excluding infectious pneumonia
  * Skin toxicity
  * Hemoptysis/pulmonary hemorrhage
  Grade 5 toxicities, including:
  * Pulmonary toxicity including pneumonitis
  * Excluding infectious pneumonia
  Three participants will enter the study in each cohort. If 0/3 patients experiences a DLT, this dose level will move forward to the Phase II and more participants will be enrolled.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Dose Level 2 [Phase I]
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Overall Response Rate [Phase II]
Description: Percentage of participants with response after 6 weeks. Response on treatment was considered to be Complete Response (CR) and Partial Response (PR) measured according Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. For target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter.
Time Frame: 6 weeks
Population: It is pre-specified in the protocol that Phase I and Phase II populations for each cohort are combined for this analysis
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 Dose Level 2 [Phase I and II]
Number analyzed (Participants) | 5
percentage of participants | 100 [54.9 to 100]

3. Secondary Outcome: Complete Response Rate [Phase II]
Description: Percentage of pulmonary lesions of participants with response after 6 weeks. Response on treatment was considered to be Complete Response (CR) measured according Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. For target lesions, CR is complete disappearance of all target lesions.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of pulmonary lesions
Units Other Than Participants: lesions
Arm/Group | Cohort 2 Dose Level 2 [Phase I and II]
Number analyzed (Participants) | 5
Number analyzed (lesions) | 8
percentage of pulmonary lesions | 75 [39 to 100]

4. Secondary Outcome: 2 Year Local Control Rate [Phase II]
Description: Rate of local control (LC) of the index lesion after lung SBRT at 2 years. LC is defined as the absence of tumor progression within 1 cm of the primary tumor site. LC is measured by established methods.
Time Frame: 24 Months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of pulmonary lesions
Units Other Than Participants: Lesions
Arm/Group | Cohort 2 Dose Level 2 [Phase I and II]
Number analyzed (Participants) | 5
Number analyzed (Lesions) | 8
percentage of pulmonary lesions | 60 [19 to 100]

5. Secondary Outcome: Percentage of Participants With 2-Year Failure-Free Survival [Phase II]
Description: Rate of distant lung failure-free survival defined lung failure or death from any cause at two years. Lung failure defined using established methods.
Time Frame: 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 Dose Level 2 [Phase I and II]
Number analyzed (Participants) | 5
percentage of participants | 40 [0 to 100]

6. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events [Phase I and II]
Description: Grade 3 or higher adverse events as defined by controlled terminology criteria for adverse events (CTCAE) version 4.
Time Frame: Up to 6 months post-treatment (6 months and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Dose Level 2 [Phase I] | Cohort 2 Dose Level 2 [Phase II]
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months post-treatment (6 months and 2 weeks)
Description: Serious Adverse Events (SAE's) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Cohort 2 Dose Level 2 [Phase I] | Cohort 2 Dose Level 2 [Phase II]
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2 Dose Level 2 [Phase I] (N=3) | Cohort 2 Dose Level 2 [Phase II] (N=2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study had small sample size / weak accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT02581384/Prot_SAP_000.pdf